CLINICAL TRIAL: NCT00159679
Title: A 13 Week, Double-Blind, Placebo-Controlled Phase 4 Trial of Pregabalin (CI-1008, 600 mg/Day) for Relief of Pain in Subjects With Painful Diabetic Peripheral Neuropathy
Brief Title: Pregabalin in the Treatment of Pain Due to Diabetic Peripheral Neuropathy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A0081060
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2021-01-25 (Actual); Status verified 2009-04

CONDITIONS: Diabetic Neuropathy, Painful
MeSH Terms: conditions — Diabetic Neuropathies | interventions — Pregabalin

INTERVENTIONS:
Drug: Pregabalin

SUMMARY:
The purposes of this study are to: 1) find out if pregabalin relieves pain in subjects with painful diabetic peripheral neuropathy; 2) find out if pregabalin is safe at a dose of 600 mg/day (taken twice a day); and 3) find out if changes in nerve function happen during the study.

ELIGIBILITY:
Inclusion Criteria:

* Adults with Type 1 or 2 diabetes
* Patients must have pain in their lower legs or feet due to painful diabetic neuropathy that has lasted for at least 3 months

Exclusion Criteria:

* Patients must not be in poor or unstable health.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2004-09; Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Nerve conduction measurements; Pain scores from patient diaries

SECONDARY OUTCOMES:
Proportion of patients with at least a 50% reduction in pain scores; Short-Form McGill Pain Questionnaire; Sleep interference scores from patient diaries; Clinical Global Impression of Change; Patient Global Impression of Change

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (22):
- United States (22):
  - Pfizer Investigational Site, Hot Springs, Arkansas
  - Pfizer Investigational Site, La Jolla, California
  - Pfizer Investigational Site, Torrance, California
  - Pfizer Investigational Site, Denver, Colorado
  - Pfizer Investigational Site, Lake Worth, Florida
  - Pfizer Investigational Site, Ocala, Florida
  - Pfizer Investigational Site, Palm Beach Gardens, Florida
  - Pfizer Investigational Site, Sunrise, Florida
  - Pfizer Investigational Site, West Palm Beach, Florida
  - Pfizer Investigational Site, Boston, Massachusetts
  - Pfizer Investigational Site, Omaha, Nebraska
  - Pfizer Investigational Site, Las Vegas, Nevada
  - Pfizer Investigational Site, Englewood, New Jersey
  - Pfizer Investigational Site, New Brunswick, New Jersey
  - Pfizer Investigational Site, Albany, New York
  - Pfizer Investigational Site, Rochester, New York
  - Pfizer Investigational Site, Greenville, North Carolina
  - Pfizer Investigational Site, Toledo, Ohio
  - Pfizer Investigational Site, Duncansville, Pennsylvania
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, San Antonio, Texas

REFERENCES:
- [Derived] Alexander J Jr, Edwards RA, Manca L, Grugni R, Bonfanti G, Emir B, Whalen E, Watt S, Brodsky M, Parsons B. Integrating Machine Learning With Microsimulation to Classify Hypothetical, Novel Patients for Predicting Pregabalin Treatment Response Based on Observational and Randomized Data in Patients With Painful Diabetic Peripheral Neuropathy. Pragmat Obs Res. 2019 Oct 31;10:67-76. doi: 10.2147/POR.S214412. eCollection 2019. PMID 31802967
- [Derived] Alexander J Jr, Edwards RA, Brodsky M, Manca L, Grugni R, Savoldelli A, Bonfanti G, Emir B, Whalen E, Watt S, Parsons B. Using time series analysis approaches for improved prediction of pain outcomes in subgroups of patients with painful diabetic peripheral neuropathy. PLoS One. 2018 Dec 6;13(12):e0207120. doi: 10.1371/journal.pone.0207120. eCollection 2018. PMID 30521533
- [Derived] Edwards RA, Bonfanti G, Grugni R, Manca L, Parsons B, Alexander J. Predicting Responses to Pregabalin for Painful Diabetic Peripheral Neuropathy Based on Trajectory-Focused Patient Profiles Derived from the First 4 Weeks of Treatment. Adv Ther. 2018 Oct;35(10):1585-1597. doi: 10.1007/s12325-018-0780-3. Epub 2018 Sep 11. PMID 30206821
- [Derived] Parsons B, Li C, Emir B, Vinik AI. The efficacy of pregabalin for treating pain associated with diabetic peripheral neuropathy in subjects with type 1 or type 2 diabetes mellitus. Curr Med Res Opin. 2018 Nov;34(11):2015-2022. doi: 10.1080/03007995.2018.1509304. Epub 2018 Sep 20. PMID 30084288
- [Derived] Markman JD, Jensen TS, Semel D, Li C, Parsons B, Behar R, Sadosky AB. Effects of Pregabalin in Patients with Neuropathic Pain Previously Treated with Gabapentin: A Pooled Analysis of Parallel-Group, Randomized, Placebo-controlled Clinical Trials. Pain Pract. 2017 Jul;17(6):718-728. doi: 10.1111/papr.12516. Epub 2016 Dec 1. PMID 27611736
- [Derived] Arezzo JC, Rosenstock J, Lamoreaux L, Pauer L. Efficacy and safety of pregabalin 600 mg/d for treating painful diabetic peripheral neuropathy: a double-blind placebo-controlled trial. BMC Neurol. 2008 Sep 16;8:33. doi: 10.1186/1471-2377-8-33. PMID 18796160